CLINICAL TRIAL: NCT07238413
Title: Investigation of the Effect of Scapular Stabilization Exercises Applied in Addition to Extracorporeal Shock Wave Therapy on Pain, Muscle Strength, Functional Status, and Quality of Life in Patients With Lateral Epicondylitis
Brief Title: Effect of Scapular Stabilization Exercises and ESWT in Patients With Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Büşra Yalçın, MSc Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TR ISTANBU60
Record Dates: First submitted 2025-09-28; First posted 2025-11-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: tennis elbow; ESWT; Pain; Scapular muscle training; functional status
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Study model
Who Masked: Outcomes Assessor
Masking Description: Masking was applied at the outcome assessment level. The independent outcome assessor was blinded to participants' group allocation throughout data collection, ensuring unbiased evaluation of study endpoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Participants in the control group will receive a protocol consisting of extracorporeal shock wave therapy (ESWT), stretching exercises for the extensor carpi radialis brevis (ECRB) muscle and wrist extensor muscles, as well as isometric, eccentric, and concentric strengthening exercises targeting the wrist extensors.
  The ESWT will be applied once a week, for a total of 5 sessions
  Interventions: Other: ESWT + Scapular stabilization exercise program
- Study group (Experimental): Participants in the study group will follow a treatment protocol consisting of extracorporeal shock wave therapy (ESWT) - 5 sessions, once per week - combined with stretching exercises for the extensor carpi radialis brevis (ECRB) and wrist extensor muscles, strengthening exercises for the wrist extensors, and an additional scapular stabilization exercise program. This combined program will be performed twice per week for a duration of 8 weeks.
  The scapular stabilization component will include strengthening exercises targeting the lower and middle trapezius and serratus anterior muscles. The program will consist of scapular clock exercises, wall push-up exercises, and wall slide or ball slide exercises performed on a wall.
  Interventions: Other: ESWT + Scapular stabilization exercise program

INTERVENTIONS:
Other: ESWT + Scapular stabilization exercise program — Participants in the study group will follow a treatment protocol consisting of extracorporeal shock wave therapy (ESWT) - 5 sessions, once per week - combined with stretching exercises for the extensor carpi radialis brevis (ECRB) and wrist extensor muscles, strengthening exercises for the wrist extensors, and an additional scapular stabilization exercise program. This combined program will be performed twice per week for a duration of 8 weeks.
  The scapular stabilization component will include strengthening exercises targeting the lower and middle trapezius and serratus anterior muscles. The program will consist of scapular clock exercises, wall push-up exercises, and wall slide or ball slide exercises performed on a wall.

SUMMARY:
We aim to investigate the effects of adding scapular stabilization exercises to the extracorporeal shock wave therapy (ESWT) protocol in the treatment of lateral epicondylitis on pain, muscle strength, functional status, and quality of life.

DETAILED DESCRIPTION:
Forty eight volunteer participants with lateral epycondilitis aged 18 to 65 years were included in the study. Participants were randomly divided into two groups as study and control group. In the control group, a protocol including ESWT, stretching of the ECRB muscle and wrist extensor muscles, and isometric, eccentric, and concentric strengthening exercises for the wrist extensors will be applied.

In the study group, the same protocol will be administered (ESWT, stretching of the ECRB and wrist extensor muscles, and strengthening exercises), with the addition of scapular stabilization exercises.

The exercise program will be conducted twice a week for 8 weeks. At the beginning of the treatment and at the end of the eighth week, pain, muscle strength, functional status, and Quality of Life were evaluated between groups

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.

  * Diagnosed with lateral epicondylitis by a physician, with positive Mill's, Cozen's, or Thomsen tests.
  * Experiencing pain and tenderness over and around the lateral epicondyle for at least 3 months, with symptoms exacerbated by resisted elbow extension, wrist extension, gripping, and supination.
  * Willing to voluntarily participate in the study.

Exclusion Criteria:

* • Individuals with serious systemic or cardiovascular diseases that contraindicate exercise of the hand and upper extremity.

  * Those diagnosed with upper extremity entrapment neuropathies.
  * Patients with a diagnosis of malignancy.
  * Individuals with open wounds on the hand or upper extremity.
  * Pregnant women or those suspected of being pregnant.
  * Patients who have received physiotherapy and/or injection treatments within the last 6 weeks.
  * Patients with diabetes mellitus, rheumatologic diseases, or neurological disorders.
  * Individuals who have undergone upper extremity surgery or had an upper extremity fracture within the last 6 months.
  * Patients with coagulation disorders or those receiving anticoagulant therapy.
  * Individuals with conditions causing degenerative changes in the hand and upper extremity.
  * Patients diagnosed with carpal tunnel syndrome, cubital tunnel syndrome, thoracic outlet syndrome, medial epicondylitis, radiohumeral bursitis, or cervical disc pathology.
  * Patients using analgesic or anti-inflammatory medications other than acetaminophen (paracetamol).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment: Visual Analog Scale (VAS) | From baseline assesment to the end of treatment at 8 weeks
  Pain will be assessed using the Visual Analog Scale (VAS). On this scale, a score of 0 indicates "no pain" and a score of 10 represents "the worst possible pain." Participants will be asked to mark their perceived pain level on a 10 cm horizontal line, anchored at 0 and 10. The distance from the left end of the line to the participant's mark will be measured in centimeters and recorded. The VAS is a valid and reliable tool for pain assessment. Pain will be evaluated separately at rest, during activity, and at night.
Scapular Position Assessment: (Lateral Scapular Slide Test) | From enrollment to the end of treatment at 8 weeks
  The distance between the inferior angle of each scapula and the nearest spinous process will be measured in three different test positions on both sides using a measuring tape.
  A side-to-side difference of 1.5 cm or more is considered a positive result and indicates scapular asymmetry.
Pressure Pain Threshold Measurement | From enrollment to the end of treatment at 8 weeks
  Measurements will be performed with a digital algometer while the participant is seated, with the shoulder abducted at 30°, the elbow flexed at 90°, and the forearm, wrist, and hand supported. Pressure pain threshold will be measured over the lateral epicondyle. Three measurements will be taken at each point using the 1 cm² tip of the algometer, and the average of these three measurements will be recorded.
Grip Strength | From enrollment to the end of treatment at 8 weeks
  Patients' grip strength will be assessed using a Jamar hand dynamometer, following the protocol recommended by the American Society of Hand Therapists.
Muscle Strength | 0 and 8 week
  Muscle strength of the lower and middle trapezius, serratus anterior, and wrist extensor muscles will be measured using a handheld dynamometer before and after the treatment.
Functional Status | From enrollment to the end of treatment at 8 weeks
  PRTEE (Patient-Rated Tennis Elbow Evaluation):
  The PRTEE is designed specifically for lateral epicondylitis and consists of 15 items divided into 3 subscales. Each item is scored from 0 to 10. Higher scores on the scale indicate worse functional status.
  (The subscales assess pain, specific activities, and general daily activities.)
  JHand:
  JHand evaluates the functional status of the upper extremity and consists of 25 items. Each item is scored on a scale from 0 (no difficulty) to 4 (unable to perform). Higher scores on this scale also indicate worse functional status.

OTHER OUTCOMES:
Health-Related Quality of Life | baseline and at the end of the 8-week intervention period.
  Short Form-12 Health Survey (SF-12) is a validated and reliable questionnaire used to assess health-related quality of life. It includes 12 items covering both physical and mental health domains, and provides two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Higher scores indicate better perceived health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Büşra Yalçın, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No